CLINICAL TRIAL: NCT05231096
Title: Comparison of the Effect of Gingival Massage of Aloe-vera Gel and Sidr Honey on Chronic Periodontitis. a Randomized Clinical Trial
Brief Title: Comparison of the Effect of Gingival Massage of Aloe-vera Gel and Sidr Honey on Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Fizza Khalid, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30071991
Record Dates: First submitted 2022-01-04; First posted 2022-02-09 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Gingival Massage; Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Aloe vera gel

STUDY DESIGN:
Intervention Model Description: 105 patients with chronic periodontitis were selected in this single-blinded Randomized control clinical trial. At recruitment non-surgical therapy i-e scaling and root debridement was performed. At baseline all clinical parameters, gingival index, plaque index, bleeding on probing and pocket depths were recorded. All the participants were then randomly divided in three groups, Group A: SRD & Gingival massage with Aloe-vera gel, Group B: SRD & Gingival massage with Sidr honey and Group C SRD only. On 30th day of trial all the patients were re-examined for all the clinical parameters.
Who Masked: Outcomes Assessor
Masking Description: The individual who evaluates the outcomes was masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: SRD & Gingival massage with Aloe-vera gel. (Experimental): Group A: Scaling and Root Debridement & Gingival massage with Aloe-vera gel.
  Interventions: Other: Aloe-vera gel; Procedure: Scaling ans root Debridement
- Group B: SRD & Gingival massage with Sidr honey (Experimental): Group B: Scaling and Root Debridement & Gingival massage with Sidr honey
  Interventions: Other: sidr honey; Procedure: Scaling ans root Debridement
- Group C SRD only. (Other): Group C Scaling and Root Debridement only.
  Interventions: Procedure: Scaling ans root Debridement

INTERVENTIONS:
Other: Aloe-vera gel — Aloe-Vera gel Production Aloe vera gel used in this study was 98% aloe vera gel concentration and 2% normal saline. Preparation of aloe-vera gel consists of ripen leaf of aloe vera.(26) Aloe vera leaf was washed thoroughly under water and then cut from the center and the seeping gel was collected in sterile container and was stored at 4°C until the time of application. In our research this pure Aloe vera gel was extracted by The Pakistan Council of Scientific & Industrial Research (PCSIR) laboratory.
  Arms: Group A: SRD & Gingival massage with Aloe-vera gel.
Other: sidr honey — Honey collection Sidr (Beri) honey was used in this study. Honey was thick, raw and cold extracted from remote Pakistan afghan tribal forest belt of Sidr trees. It was smooth, viscous and medium to dark amber in color.
  Arms: Group B: SRD & Gingival massage with Sidr honey
Procedure: Scaling ans root Debridement — non-surgical periodontal therapy was given to all the participants of all the three groups

SUMMARY:
Chronic Periodontitis is an inflammatory condition and a common disease worldwide. Honey has been used in dentistry for its beneficial properties. It has been used in many oral conditions like gingivitis and periodontal diseases for its antibacterial and healing properties, on the other hand, aloe vera gel is known for its anti-inflammatory aspects, and it has been used in dentistry for its potential advantages.

Objective The main objective of the study was to find out the effects of gingival massage with aloe-vera gel and sidr honey as adjunct to non surgical therapy after one month in patients with Chronic periodontitis and to find out whether there is a difference in the efficacy of aloe-vera gel and sidr honey in reducing plaque index, gingival index, pocket depth and bleeding on probing after one month of gingival massage when used as adjunct to non-surgical therapy.

Method 105 patients with chronic periodontitis were selected in this single-blinded Randomized control clinical trial. At recruitment non-surgical therapy i-e scaling and root debridement was performed. At baseline all clinical parameters, gingival index, plaque index, bleeding on probing and pocket depths were recorded. All the participants were then randomly divided in three groups, Group A: SRD & Gingival massage with Aloe-vera gel, Group B: SRD & Gingival massage with Sidr honey and Group C SRD only. On 30th day of trial all the patients were re-examined for all the clinical parameters.

Statistical Analysis SPSS version 21 was used for data entry and analysis with significance level set at Ƥ <0.05. Median, median difference and Inter Quartile ranges were reported for plaque index, gingival index, probing depth and percentages were reported for bleeding on probing. Wilcoxon Signed rank test was used for pre and post comparison. Mann Whitney test was applied for comparison between groups.

DETAILED DESCRIPTION:
Study Design The study is a Randomized controlled clinical trial. 3.2 Study Setting The study was carried out in the department of Periodontology at Dr.Ishrat-ul-Ebad Khan Institute of Oral Health Sciences.

3.3 Study Duration The duration of the study was 6-8 months after the synopsis approval. 3.4 Study Population The study was conducted on patients with Chronic Periodontitis. 3.4.1 Inclusion Criteria

1. Male/ female, 35-65 years of age with minimal 5 natural teeth in each quadrant excluding 3rd molars.
2. Patients having Chronic Periodontitis with probing depth 4 to 6mm and bleeding on probing in 20 sites.
3. Systematically healthy individuals with Chronic Periodontitis. 3.4.2 Exclusion Criteria

1. Individuals who smoke. 2. Any addiction of Areca nuts, gutka, paan or alcohol. 3. Individuals with any systemic diseases like diabetes mellitus, cardiovascular, endocrine as they may affect the outcome of research.

4. Women with pregnancy/lactation. 5. Individuals with any known allergy from aloe-vera or honey. 6. Systemic or topical use of antibiotic in past 6 months. 3.5 Sample Size Total of 105 patients were calculated (35 in each group) by using PASS V-11, Pair sample T-test with 95% Confidence Interval and 80% Power of test. Difference of plaque index at base line versus after 1 month mean (20.02) and standard deviation (68.16). Calculated sample size is 93, which is increased to 105.(26) 3.6 Sampling Technique The sampling technique was Non Probability consecutive sampling. 3.7 Data Collection Procedure Patients attending the Department of Periodontology were approached and examined for chronic periodontitis. Patients with chronic periodontitis were explained the research study procedure. Patient signing the consent form was enrolled in the study. All the enrolled participants went through a detailed history which includes medical health, systemic illness, regular medications, hospitalizations, any known allergies, dental checkups, any bad oral habit and routine oral hygiene practice. Any entrant having any allergy from honey or aloe-vera gel or anyone falling in our exclusion criteria were not selected in our research. All those who fulfilled our criteria were clinically examined and all the clinical parameters were recorded by the principal investigator at the baseline, i-e, pocket depth, gingival index, plaque index and bleeding on probing. Probing depth was recorded by Goldman-Fox probe with William's markings and flattened surface. Probing depth measurement was done by inserting probe on six sites on each tooth (mesial, distal, mid lingual, mid buccal, buccal and lingual), all the markings were measured from the marginal gingiva to the base of the periodontal pocket and were recorded in millimeters, if the tooth has recession and clinical attachment loss in any site of tooth it was not measured and was not included in our study. Bleeding on probing was checked on the buccal and lingual sulcus of tooth after inserting the probe and wait for 30 seconds, if bleeding occurs bleeding on probing was considered as 1 and labeled as positive bleeding on probing and if there is no bleeding it was considered as 0 and labeled as no bleeding on probing, Percentage of BOP was recorded by dividing positive bleeding sites by total number of sites present in each patient multiplied by 100. Gingival index (Loe and Silness, 1963) were recorded as score 0: Normal gingiva, 1: Mild inflammation on gingiva, 2: Moderate inflammation on gingiva and 3: Severe inflammation on gingiva. Plaque index (Loe and Silness, 1964) was recorded as score 0: No plaque, 1: plaque film on free gingival margin, 2: Moderate plaque on gingival margin; can be seen by the naked eye, 3: Abundance of soft matter in gingival pocket. After recording all the clinical parameters principal investigator performed non-surgical therapy (scaling and root debridement) by using ultrasonic scalers in single visit. Following scaling and root debridement the participants of all the three groups were given detailed oral hygiene instructions with demonstration of proper brushing technique i-e Modified Bass technique. After that all the participants were provided with a regular cleaning kit which consist of fluoride toothpaste (Colgate® Cavity Protection Toothpaste) and toothbrush (Colgate® Classic Clean Toothbrush) Moreover, all enrolled patients in Group A and B were minutely demonstrated by principal investigator for gingival massage.

Aloe-Vera gel Production Aloe vera gel used in this study was 98% aloe vera gel concentration and 2% normal saline. Preparation of aloe-vera gel consists of ripen leaf of aloe vera.(26) Aloe vera leaf was washed thoroughly under water and then cut from the center and the seeping gel was collected in sterile container and was stored at 4°C until the time of application. In our research this pure Aloe vera gel was extracted by The Pakistan Council of Scientific & Industrial Research (PCSIR) laboratory.

Honey collection Sidr (Beri) honey was used in this study. Honey was thick, raw and cold extracted from remote Pakistan afghan tribal forest belt of Sidr trees. It was smooth, viscous and medium to dark amber in color.

Random Allocation of the Intervention A total of 105 participants were divided in to three groups and were named as Group A: SRD & Gingival massage with Aloe-Vera gel, Group B: SRD & Gingival massage with Sidr honey and group C: SRD only. Interventions were randomly allocated. For this purpose, entrants were asked to pick one sealed opaque envelope in which random allocation of the interventions were mentioned. All the participants who were in Group A and B were not blinded and trained for gingival massage by principal investigator. All the participants were guided to rub aloe-vera gel or sidr honey on the skin of wrist first to recheck any allergy. At last participants were trained for application of the material gently on the gingiva and the gingival sulcus of all the teeth. To perform gingival massage patients used the index finger of their dominant hand, applied the material at the bottom of their gums with slight pressure, then moved the finger in a slow and circular motion/rubbing action for 1 to 3 minutes, after performing the massage patients were not allowed to rinse with water or any other fluids for 30 minutes for further retaining the material on the gingiva and in the gingival sulcus thereby preventing washing out of the material. All the patients were instructed to perform gingival massage with aloe-vera gel and sidr honey twice a day after meals and to wait for 30 minutes after application of the interventions. All the routine oral hygiene practice which includes brushing twice a day (morning and night) was continued as usual. Patients falling in the control group were instructed to follow routine oral hygiene protocols. Telephonic communications were made weekly for encouraging the patients for gingival massage with given interventions. All the patients were recalled on 30th day for Post-intervention assessment. The baseline clinical parameters were recorded by principal investigator whereas 1 month follow-up of all clinical parameters were recorded by a trained examiner in this study. Intra-examiner reliability was checked to ensure calibration between examiners. For this purpose both examiners recorded clinical parameters of 50 subjects with chronic periodontitis who were not involved in our study and reliability came out to be 88%. The trained examiner who was blinded from the intervention given to patients was asked to re-assess all the clinical parameters which included periodontal pocket depth, gingival index, plaque index and bleeding on probing.

ELIGIBILITY:
Inclusion Criteria

* Male/ female, 35-65 years of age with minimal 5 natural teeth in each quadrant excluding 3rd molars.
* Patients having Chronic Periodontitis with probing depth ≥ 4 to 6mm and bleeding on probing in greater than 20% sites.
* Systematically healthy.

Exclusion Criteria:

* Individuals who smoke.
* Any addiction of Areca nuts, gutka, paan or alcohol.
* Individuals with any systemic diseases like diabetes mellitus, cardiovascular, endocrine as they may affect the outcome of research.
* Women with pregnancy/lactation.
* Individuals with any known allergy from aloe-vera or honey.
* Systemic or topical use of antibiotic in past 6 months.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Periodontal pocket depth | 1 month
  pocket depths were measured on tooth and probing depths with 4-6mm were included.
Gingival index | 1 month
  Score 0=Normal gingiva Score 03=Severe inflammation - marked redness and edema. Ulceration. Tendency to spontaneous bleeding.
Plaque index | 1 month
  Score 0=No plaque in the gingival area. Score 03=Abundance of soft matter within the gingival pocket or on gingival margin
Bleeding on probing. | 1 month
  recorded on each tooth and greater than 20% bleeding on probing sites were selected.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Fizza, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Khalid F, Ahmed S, Farooqui WA, Pervaiz H, Riaz S, Shabbir S, Ghazal M, Khan ZR. Clinical Assessment of the Efficacy of Natural Nutraceuticals in Gingival Massage Therapy: A Randomized Clinical Study. Int J Dent Hyg. 2025 Dec 10. doi: 10.1111/idh.70014. Online ahead of print. PMID 41373073